CLINICAL TRIAL: NCT03098472
Title: Cholinesterase Activity and Delirium During Critical Illness Study
Acronym: CADUCeuS
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: DR. FRANZ KOHLER CHEMIE GMBH (Unknown)
Responsible Party: Principal Investigator, Christopher G Hughes, Associate Professor of Anesthesiology, Vanderbilt University Medical Center
Other Study IDs: CADUCeuS
Record Dates: First submitted 2017-03-22; First posted 2017-03-31 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Delirium; Cognitive Impairment
MeSH Terms: conditions — Delirium; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Delirium is a syndrome of acute brain dysfunction involving attention and cognition that affects up to half of older hospitalized patients and 50%-75% of critically ill ICU patients, such that millions of patients worldwide experience this acute threat to their health and well being every year. One-third to half of critical illness survivors struggle with a dementia-like disorder similar in severity to moderate-to-severe traumatic brain injury or Alzheimer's Disease, and the only proven risk factor that is potentially modifiable is delirium in the ICU. Despite the frequency and impact of delirium in the ICU, little is known regarding the biological mechanisms that lead to this form of organ dysfunction during critical illness. A widely held hypothesis proposes that inflammation is regulated by the cholinergic system, and that this interaction plays a pivotal role whether delirium developments in the setting of acute illness. Acetylcholinesterase (AChE) and butyrylcholinesterase (BuChE) are enzymes that hydrolyze the neurotransmitter acetylcholine. Changes in the activity of these enzymes, which can be measured in whole blood, reflect altered regulation of circulating acetylcholine. AChE and BuChE activities have promise as both predictors of delirium (when found to be low at admission) and biomarkers of delirium (when low during serial measurement). Neither of these biomarkers, however, have been studied in the ICU setting where delirium risk is the highest. The current investigation, therefore will be the first to determine the validity of circulating AChE and BuChE activities as biomarkers of delirium during critical illness and subsequent cognitive impairment after discharge. This study will measure whole blood AChE and butyrylcholinesterase BuChE activities within the framework of the ICU Delirium and Cognitive Impairment Study Group's ongoing clinical trials in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults (>18 years of age) treated for acute respiratory failure (with mechanical ventilation or non-invasive positive pressure ventilation [NIPPV]) and/or shock (with vasopressors) in a medical and/or surgical ICU at Vanderbilt University Medical Center enrolled in an ICU Delirium and Cognitive Impairment Study Group's clinical trials. Exclusion criteria for the parent studies are summarized below. No additional exclusion criteria are required for this investigation.

Exclusion Criteria:

* Expected death within 24 hours of enrollment or lack of commitment to aggressive treatment by family or the medical team (e.g., likely withdrawal of life support measures within 24 hours of screening)
* Active substance abuse, psychotic disorder, or homelessness without a secondary contact person (which would make long-term follow-up difficult)
* Blindness or deafness (which would prevent assessment of the study's outcomes)
* Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include all patients in the ICU Delirium and Cognitive Impairment Study Group's ongoing clinical trials over a two-year period of time.
Sampling Method: Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Delirium | During hospital stay until death or hospital discharge, whichever comes first, up to 30 days
  Confusion Assessment Method for the ICU

SECONDARY OUTCOMES:
Global cognition | At 3, 6, and/or 12 months after hospital discharge up to 18 months after discharge
  Neuropsychological battery

OTHER OUTCOMES:
Activities of daily living | At 3, 6, and/or 12 months after hospital discharge up to 18 months after discharge
  Katz Index of Independence in Activities of Daily Living
Instrumental activities of daily living | At 3, 6, and/or 12 months after hospital discharge up to 18 months after discharge
  Functional activities questionnaire
Quality of life and generic health status | At 3, 6, and/or 12 months after hospital discharge up to 18 months after discharge
  EQ-5D
Coma | During hospital stay until death or hospital discharge, whichever comes first, up to 30 days
  Richmond Agitation Sedation Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hughes CG, Boncyk CS, Fedeles B, Pandharipande PP, Chen W, Patel MB, Brummel NE, Jackson JC, Raman R, Ely EW, Girard TD. Association between cholinesterase activity and critical illness brain dysfunction. Crit Care. 2022 Dec 6;26(1):377. doi: 10.1186/s13054-022-04260-1. PMID 36474266